CLINICAL TRIAL: NCT02598258
Title: Hemodynamic Effects of Dry Sauna Followed by Cold Water Immersion in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Mathieu Gayda, Professeur agrégé de clinique, Montreal Heart Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 15-1807
Record Dates: First submitted 2015-10-08; First posted 2015-11-05 (Estimated); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Blood Pressure; Arrhythmias
Keywords: Sauna; Cold water bath
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Steam Bath

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sauna + Cold Water Bath (Experimental): Subjects will first spend 10 minutes in a dry sauna at 85 degrees celtius. Immediately after , subjects will be immersed in a cold water bath (ICool , Australia) at a temperature of 5 degrees celtius for approximately one minute. Blood pressure , ecg , gaz exchange and thoracic impedance will be measured during sauna and cold water bath.
  Interventions: Other: Sauna and cold water bath

INTERVENTIONS:
Other: Sauna and cold water bath — Subjects will first spend 10 minutes in a dry sauna at 85 degrees celtius. Immediately after, subjects will be immersed in a cold water bath (ICool , Australia) at a temperature of 5 degrees celtius for approximately one minute. Blood pressure , ecg , gaz exchange and thoracic impedance will be measured during sauna and cold water bath.

SUMMARY:
The purpose of this study is to determine the safety on sauna followed by cold water bath, a common practice in many countries, 30 healthy subjects aged 40 years and older will be at the Montreal Heart Institute Prevention and Cardiac Rehabilitation centre.

DETAILED DESCRIPTION:
To determine the safety on sauna followed by cold water bath, a common practice in many countries, 30 healthy subjects aged 40 years and older will be at the Montreal Heart Institute Prevention and Cardiac Rehabilitation centre. A recent complete evaluation will have excluded any cardiac condition. Subjects will first spend 10 minutes in a dry sauna at 85 degrees celtius. Immediately after , subjects will be immersed in a cold water bath (ICool , Australia) at a temperature of 5 degrees celtius for approximately one minute. Blood pressure , ecg , gaz exchange and thoracic impedance will be measured during sauna and cold water bath.

Principal goal of study: to determine the safety of this practice. Secondary goals of study: to measure the blood pressure response, heart rate, presence of arrythmyas, cardiac output and cerebral perfusion during both conditions.

Primary endpoint: Change in systolic blood pressure from sauna (after 10 minutes ) to cold water (after one minute).

Physiologic measurements: continuous ECG monitoring, BP measurements at every 3 minutes during sauna and at one minute in the cold bath, gaz exchange with a portable equipment (Cosmed K4), bioimpedance and cerebral perfusion with a single frontal NIRS electrode.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women and men aged 40 and older with a recent complete medical evaluation including a normal resting ECG and a normal symptom-limited treadmill exercise test.

Exclusion Criteria:

* Any cardiac condition, abnormal exercise test, hypertension, type I diabetes and presence of any medications that may affect blood pressure.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Blood pressure | Difference between baseline and 11 minutes of intervention.

SECONDARY OUTCOMES:
Arrhytmias | Number of arrhytmias during all 25 minutes of the intervention.
  Patients will use a HOLTER during all experiment. Total time: 25 minutes.
Blood pressure | Measured at 10 minutes after the end of the intervention (recovery period).

CONTACTS AND LOCATIONS:
Overall Officials: Martin Juneau, Principal Investigator — EPIC Centrer - Montreal Heart Institute
Locations (1):
- Cardiovascular Prevention and Rehabilitation Center, Montreal, Quebec, Canada